CLINICAL TRIAL: NCT06669338
Title: The Effect of Music Therapy and White Noise on Pre-procedural Fear, Anxiety and Vital Signs of Elderly Colonoscopy Patients: A Double-Blind Randomized Controlled Trial
Brief Title: Effects of Music Therapy and White Noise on Pre-procedural Fear, Anxiety by Elderly Colonoscopy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Mehtap Cullu, Phd lecturer, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MuglaSKU-HEM-MC-01
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Colonoscopy; the Elderly; White Noise; Music Therapy; Fear; Anxiety
Keywords: Colonoscopy;anxiety;fear;vital signs;musictherapy;whitenoise
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: experimental study with three groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: results evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- music therapy group (Experimental): The group that listened to music for 20 minutes before the colonoscopy
  Interventions: Other: Music therapy
- white noise group (Experimental): The group that listened to white noise for 20 minutes before the colonoscopy
  Interventions: Other: listen to white noise
- control group (Placebo Comparator): The group that listened to recorded ambient sound for 20 minutes before the colonoscopy.
  Interventions: Other: listen to hospital ambient sound

INTERVENTIONS:
Other: Music therapy — patients listen to music for 20 minutes with headphones before colonoscopy.
  Arms: music therapy group
Other: listen to white noise — patients listen to white noise with headphones for 20 minutes before colonoscopy.
  Arms: white noise group
Other: listen to hospital ambient sound — patients listen to recorded ambient sound for 20 minutes with headphones before colonoscopy.
  Arms: control group

SUMMARY:
The aim of the study was to examine the effect of two different interventions (music therapy and white noise listening) on anxiety, fear and vital signs in elderly patients undergoing colonoscopy.

The study was a double-blind, pre-test and post-test

DETAILED DESCRIPTION:
Colonoscopy patients experience high levels of fear and anxiety due to the procedure. Fear and anxiety can activate the patient's autonomic nervous system, leading to increased sweating, increased heart rate, blood pressure and respiratory rate, and procedure-related complications. Reducing fear and anxiety and relaxing the patient not only prevents potential harm to the patient due to the procedure, but also facilitates the work of the healthcare team performing the procedure and ensures accurate results. In this context, this study aimed to investigate the effects of music therapy and white noise listening on the fear, anxiety and vital signs of patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. The one to be colonoscoped,
2. 65 years of age or older,
3. Participated in the research voluntarily
4. No vision, hearing and perception problems,
5. No communication problems (able to speak Turkish),
6. Those who are hemodynamically stable before colonoscopy,
7. No psychiatric diagnosis, no use of antidepressants, anxiolytics and sedative agents,
8. No analgesic or anesthetic medication 24 hours before the procedure.

Exclusion Criteria:

1. Developing complications during the procedure,
2. Removing the headset during the procedure,
3. Participants with visual and hearing impairment or a medical history of dementia, cognitive impairments or psychiatric disorders
4. The general condition deteriorated during the procedure or a different intervention was performed with anesthesia,
5. Who wants to leave the study on their own accord.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
respiratory rate | 20 minutes of music therapy, white noise and ambient sound before colonoscopy.
  Measurements are made at the beginning and end of the music therapy, white noise and ambient sound listening intervention before colonoscopy.

SECONDARY OUTCOMES:
diastolic blood pressure | 20 minutes of music therapy, white noise and ambient sound before colonoscopy.
  Measurements are made at the beginning and end of the music therapy, white noise and ambient sound listening intervention before colonoscopy.
Visual Analog Scale (VAS) | 20 minutes of music therapy, white noise and ambient sound before a colonoscopy.
  Measurements are made at the beginning and end of the music therapy, white noise and ambient sound listening intervention before colonoscopy.
The State-Trait Anxiety Inventory (STAI-I) | 20 minutes of music therapy, white noise and ambient sound before colonoscopy.
  The scale is administered before colonoscopy, at the beginning and at the end of the music therapy, white noise and ambient sound listening intervention.
heart rate | 20 minutes of music therapy, white noise and ambient sound before colonoscopy.
  Measurements are made at the beginning and end of the music therapy, white noise and ambient sound listening intervention before colonoscopy.
SpO2: peripheral oxygen saturation (%) | 20 minutes of music therapy, white noise and ambient sound before colonoscopy.
  Measurements are made at the beginning and end of the music therapy, white noise and ambient sound listening intervention before colonoscopy.
systolic blood pressure | 20 minutes of music therapy, white noise and ambient sound before colonoscopy.
  Measurements are made at the beginning and end of the music therapy, white noise and ambient sound listening intervention before colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap ÇULLU, PhD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (2):
- Turkey (Türkiye) (2):
  - Mugla, Muğla, Mentese
  - Mugla, Muğla

IPD SHARING:
Plan to Share IPD: No
Taking time to share data and not having the time to do so,
  There is no benefit in sharing data,